CLINICAL TRIAL: NCT01838187
Title: An Open Label, Expanded Access Protocol Using 131I-METAIODOBENZYLGUANIDINE (131I-MIBG) Therapy +/- Vorinostat in Patients With Refractory Neuroblastoma, Pheochromocytoma, or Paraganglioma
Brief Title: Expanded Access Protocol Using 131I-MIBG Therapy +/- Vorinostat for Refractory Neuroblastoma, Pheochromocytoma, or Paraganglioma
Status: No longer available | Type: Expanded Access
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: MIBG Expanded Access (NDP)
Record Dates: First submitted 2013-04-08; First posted 2013-04-23 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Neuroblastoma; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma; Paraganglioma | interventions — 3-Iodobenzylguanidine; Vorinostat

INTERVENTIONS:
Radiation: I-131 MIBG — The therapeutic dose (5-18 mCi/kg at investigator's discretion; any dose ≥12 mCi/kg requires stored stem cells) will be diluted in normal saline, and will be infused intravenously over 90-120 minutes.
  Other Names: ◦I-131 Iobenguane; ◦I-131 meta-iodobenzylguanidine
Drug: Vorinostat — 180 mg/m2 orally once daily on days 0 to +13
  Other Names: SAHA (suberanilohydroxamic acid); Zolinza

SUMMARY:
Currently there is no known effective treatment for patients with advanced stage neuroblastoma who have relapsed or not responded to standard therapy. There is also no known effective treatment for patients with pheochromocytoma or paraganglioma who are less than 12 years of age. In previous studies that used 131I-MIBG as a potential anti-cancer therapy, a decrease in the size of tumors was seen in some of the children and adults. This research study will continue to evaluate the side effects of 131I-MIBG +/- Vorinostat when treating children and adults with neuroblastoma, pheochromocytoma, or paraganglioma. The 131I-MIBG compound is intended to work by selectively delivering the radioactive iodine to the tumor cells, which is then intended to result in their destruction.

The purpose of this research study is to:

* Make 131I-MIBG therapy available to patients with advanced neuroblastoma, pheochromocytoma, or paraganglioma
* Further assess the side effects of 131I-MIBG therapy

DETAILED DESCRIPTION:
Neuroblastoma, pheochromocytoma, and paraganglioma remain fatal diseases for a large percentage of patients, especially those with high-risk disease features who become resistant to conventional therapy. 131I-metaiodobenzylguanidine (131I-MIBG) is a norepinephrine analog that concentrates in adrenergic tissue and has been shown to be sensitive and specific for detecting localized and metastatic neuroblastoma, pheochromocytoma, and paraganglioma. More importantly, experience of many institutions has proven that this agent used as a targeted radiotherapeutic has significant anti-tumor activity against refractory neuroblastoma 1-7 as well as pheochromocytoma and paraganglioma. Children's Hospital of Philadelphia, UCSF, and the University of Michigan have just completed a large Phase 2 study of 131I-MIBG given in doses of 10-18 mCi/kg with stem cell rescue, if necessary, and have shown that this agent is safe and effective palliative therapy for refractory or relapsed neuroblastoma patients. In addition, there is growing evidence that low-dose (5-10 mCi/kg) submyeloablative MIBG therapy is both safe and effective for disease palliation. In addition, a recently published randomized phase 2 trial in patients with relapsed/refractory neuroblastoma showed that the combination of vorinostat/MIBG had a higher response rate than 131I-MIBG alone, with manageable toxicity. This protocol therefore provides a mechanism to deliver this therapy when clinically indicated.

Primary Objectives:

* Provide palliative therapy with MIBG + vorinostat for patients with advanced neuroblastoma who can take vorinostat
* Provide palliative therapy with MIBG without vorinostat for patients with advanced neuroblastoma who cannot take vorinostat, and those with pheochromocytoma, or paraganglioma
* Gain more information about acute and late toxicity of 131I-MIBG therapy +/- vorinostat for patients with refractory neuroblastoma, and 131I-MIBG therapy alone for those with pheochromocytoma, or paraganglioma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Refractory/Relapsed neuroblastoma with original diagnosis based on tumor histopathology or elevated urine catecholamines with typical tumor cells in the bone marrow. Age ≥ 12 months and able to cooperate with radiation safety restrictions during therapy period with/without pharmacologic anxiolysis.These patients are eligible for MIBG with or without Vorinostat per investigator discretion and eligibility criteria below.
* Pheochromocytoma or paraganglioma not amendable to curative surgery. Age < 12 years and able to cooperate with radiation safety restrictions during therapy period with/without pharmacologic anxiolysis.These patients are eligible for MIBG alone.
* Disease status: Failure to respond to standard therapy (usually combination chemotherapy with/without radiation and surgery) or development of progressive disease at any time (any new lesion or an increase in size of > 25% of a pre-existing lesion). Disease evaluation must be completed within 8 weeks of study entry. If possible, the disease evaluation should take place subsequent to intervening therapy; if intervening therapy does occur, evaluations should be done as clinically indicated. If patient has received prior treatment with MIBG, they must have a response or stable disease after the most recent MIBG infusion. Patient may have PD after showing initial response to MIBG therapy (at [or around] the day 35-63 post-MIBG therapy evaluation).
* Patients must have a hematopoietic stem cell product available for re-infusion after 131I-MIBG treatment at doses of >12 mCi/kg. If no stem cells are available, then the dose of 131I-MIBG should be ≤12 mCi/kg. Vorinostat cannot be given to patients who do not have available stem cells (regardless of 131I-MIBG dose).

  * The minimum quantity for purged or unpurged peripheral blood stem cells (PBSC) is 1.5 x 10e6 viable CD34+ cells/kg (recommended 2 x 10e6 viable CD34+ cells/kg).
  * The minimum dose for bone marrow is 1.0 x 10e8 mononuclear cells/kg (optimum > 2.0 x 10e8 mononuclear cells/kg).
* Prior Therapy: Patients may enter this study with/without re-induction therapy for recurrent tumor. Patients must have fully recovered from the toxic effects of any prior therapy, meeting the following criteria: At least 2 weeks should have elapsed since any anti-tumor therapy and the patient must meet hematologic criteria below. Three-months should have elapsed in the case of completing radiation to any of the following fields: craniospinal, total abdominal, whole lung, total body irradiation (spot irradiation to skull-based metastases is NOT considered craniospinal radiation for the purposes of this study. Cytokine therapy must be discontinued a minimum of 24 hours prior to 131I-MIBG therapy.For patients who will receive vorinostat with MIBG therapy: Miniumum of four weeks since previous vorinostat. For patients who will receive vorinostat with MIBG therapy: Minimum of 7 days since taking prohibited medications that prolong QTc.
* Bilirubin ≤ 2x upper limit of normal; AST/ALT ≤ 10x upper limit of normal
* Serum Creatinine ≤ 2x upper limit of normal OR 24-hr creatinine clearance OR GFR ≥ 60 ml/min/1.73m2(For example, a patient would meet this criteria if GFR < 60 ml/min/1.73m2 but serum creatinine ≤ 2x upper limit of normal.)
* ANC ≥ 750/µL; Platelets ≥ 50,000/µL without transfusion if stem cells are not available (ANC ≥ 500 and any platelet count allowed if stem cells available). Patient must be off myeloid growth factors for at least 24 hours. If the patient has received prior treatment with MIBG, they may be thrombocytopenic, but requiring no more than 2 platelet transfusions per week to maintain counts above 20,000. Hemoglobin must be ≥ 7 gm/dL (transfusion allowed) regardless of stored stem cell availability.
* For patients who will be receiving treatment with vorinostat: PT(INR): < 1.5X ULN; PTT: <1.5X ULN
* Normal lung function as manifested by no dyspnea at rest or exercise intolerance, no oxygen requirement
* No clinically significant cardiac dysfunction
* Eligibility criteria specific for patients who will be receiving vorinostat:

  * No history of allergic reactions to vorinostat
  * No history of deep venous thrombosis (DVT)-this does not include a DVT associated with the presence of a central venous catheter
  * Patient must not be receiving prohibited medications known to prolong the QTc interval. Note this includes pentamidine, azithromycin and methadone among other medications.
  * Corrected QT (QTc) interval ≤ 480 msec
  * Has not had vorinostat toxicity requiring discontinuation of the drug previously.
* Signed informed consent/assent: The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent/assent to become a study subject has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand therapy. Significant organ impairment should be discussed with the Principal Investigator prior to patient entry.
* No patients who are pregnant or lactating will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus. Abstinence is an effective method of birth control.
* Patients who are on hemodialysis
* Proteinuria, in the absence of urinary infection, within 4 weeks prior to the planned treatment date is a relative contraindication to receiving therapy for patients with pheochromocytoma/paraganglioma. Patients with pheochromocytoma/paraganglioma with any proteinuria must have a 24-hr urine protein determination. If proteinuria is confirmed as being above the institutional upper limit of normal, the patient is ineligible for MIBG therapy.
* Patients with active infections that meet grade 3-4 according to the NCI CTCAE v5.0.
* Patients with known MIBG-avid parenchymal brain metastases are not eligible. (Patients with leptomeningeal or skull-based metastases are eligible.)
* Patients who will be receiving treatment with vorinostat: Patients receiving treatment with valproic acid and warfarin within 30 days prior to enrollment are not eligible.

Min Age: 12 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Brian Weiss, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States